CLINICAL TRIAL: NCT06163560
Title: Effectiveness of a Technology-based Developmental Guidance Program for Enhancing Infant Mental Well-being: a Randomized Controlled Trial
Brief Title: Effectiveness of a Baby App for Enhancing Infant Mental Well-being (RCT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie Wan Yee Tso (Dr), Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Babyapp_rct
Record Dates: First submitted 2023-11-20; First posted 2023-12-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Child Development
Keywords: Infant mental health; Parenting skills; Smartphone app

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Babyapp group (Experimental): This group will be provided access to the app and be asked for their feedback on the performance of the app.
  Interventions: Device: Smartphone app "Happy Baby HK"
- Control group (Active Comparator): This group will be given an information pack consisting of a parenting booklet from the Maternal and Child Health Centres (MCHC).
  Interventions: Device: Family Health Service parenting booklet

INTERVENTIONS:
Device: Smartphone app "Happy Baby HK" — "Happy Baby HK" will provide developmental stage, developmental aspects, parenting videos and cartoon images created for new mothers.
  Arms: Babyapp group
Device: Family Health Service parenting booklet — The parenting booklet is publicly available and provides brief caretaking tips for mothers with children under 3 years of age.
  Arms: Control group

SUMMARY:
This RCT aims to design and develop a developmental guidance program delivered by a smartphone app "Happy Baby HK" and evaluate its effectiveness for enhancing the mental well-being of recently born infants in Hong Kong. This study will evaluate the effectiveness of the improvement in the effect of infants and decrease of risk of developmental delay in very young children.

The smartphone app "Happy Baby HK" will be designed and developed by different professionals. Then, participants will be invited to use this app or the MCHC parenting booklet. They will also be invited to fill in some questionnaires at 6, 12 and 18 months postpartum to screen the developmental stages. Researchers will compare the intervention group and the control group to evaluate the effectiveness of this app for enhancing the mental well-being of infants.

DETAILED DESCRIPTION:
Infant mental health refers to "the developing capacity of the child from birth to age three to experience, regulate, and express emotions; form close and secure interpersonal relationships; and explore the environment and learn - all in the context of family, community, and cultural expectations for young children". Despite the stability of temperamental characteristics across context and over time, environmental factors such as good mother-infant relationship can protect against the development of psychiatric morbidities in children with difficult temperament. Research studies also show that anticipatory guidance interventions can promote optimal child development, increase maternal knowledge of their infants, positive parent-infant interactions and reduce injury rates.

To enhance infant mental well-being, the proposed project team designs a smartphone app "Happy Baby HK" that provides development guidance to mothers of recently born infants in Hong Kong. Compared to traditional approaches (e.g. parenting pamphlets or clinical consultation on developmental issues), smartphone apps devoted to parenting guidance could feature video demonstrations, quizzes, interactive games, and written information with vivid images and cartoons which are more likely to engage parents and reinforce their learning anytime and anywhere.

However, currently there is no technology-based intervention with provision of anticipatory guidance information on child development in Hong Kong.

Therefore, the objective of this study is to design and develop a developmental guidance program delivered by a smartphone app "Hapy Baby HK" and evaluate its effectiveness for enhancing the mental well-being of recently born infants in Hong Kong. The improvement on parental stress will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* mothers aged 18 years or above who attend the antenatal clinics or stay in the postnatal wards at Kwong Wah Hospital or Queen Mary Hospital at the time of recruitment and can give consent

Exclusion Criteria:

* mothers who have inability to read Chinese, no Internet access, high risk pregnancy, history of psychiatric illness,
* infants with congenital/genetic/structural abnormalities,
* infants required admission to neonatal intensive care unit

Ages: 1 Day to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 586 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
At 6 postpartum | 6 months postpatrum
  Mothers will be asked to answer the 6 months version of Ages & Stages Questionnaires.
12 months postpartum | 12 months postpatrum
  Mothers will be asked to answer the 12 months version of Ages & Stages Questionnaires.

SECONDARY OUTCOMES:
At 18 months postpartum (child development) | 18 months postpartum
  Mothers will be asked to answer the 18 months version of Ages & Stages Questionnaires.
At 18 months postpartum (screen time) | 18 months postpartum
  Mothers will be asked to answer the family questionnaire items related to child screen time use.
At 18 months postpartum (DASS-21) | 18 months postpartum
  Mothers will be asked to complete Depression Anxiety Stress Scale - 21.
At 18 months postpartum (KIDI) | 18 months postpartum
  Mothers will be asked to complete the Knowledge of Infant Development Inventory Accuracy Score.
At 18 months postpartum (PSS) | 18 months postpartum
  Mothers will be asked to complete the Parental stress scale (PSS).

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Wan Yee Tso, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Li Ka Shing Faculty of Medicine, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No